CLINICAL TRIAL: NCT06060106
Title: Endoscopic Submucosal Dissection Versus Esophagectomy for Early Esophageal Carcinoma：a Cohort Study
Brief Title: Endoscopic Submucosal Dissection Versus Esophagectomy for Early Esophageal Carcinoma
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology，Changhai Hospital；Academician of Chinese Academy of Engineering, Changhai Hospital
Other Study IDs: early esophageal carcinoma
Record Dates: First submitted 2023-06-15; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection; Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic submucosal dissection: Early esophageal cancer patients treated with ESD
  Interventions: Procedure: Endoscopic submucosal dissection
- Esophagectomy: Early esophageal cancer patients treated with esophagectomy
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — The patient was positioned in the left lateral decubitus position.Marking dots were made with a dual knife/hybrid knife around the lesion, and a solution of glycerin fructose with indigo carmine was injected into the submucosal layer to lift the lesion. Finally, after pre-cutting of the mucosal and submucosal layers around the lesion and dissection of the submucosa, the lesion was removed en bloc.
  Groups: Endoscopic submucosal dissection
Procedure: Esophagectomy — The main surgical methods of esophagectomy include the McKeown operation, Lvor-lewis, Sweet and minimally invasive radical resection of esophageal cancer (MIE)
  Groups: Esophagectomy

SUMMARY:
Endoscopic submucosal dissection (ESD) is a minimally invasive alternative to esophagectomy for early esophageal squamous cell carcinoma (EESCC), The data of EESCC patients who received ESD or esophagectomy were retrospectively analyzed,The aim of this study was to compare the efficacy and safety of ESD and esophagectomy in EESCC,Risk factors affecting the prognosis of patients with early esophageal squamous cell carcinoma were analyzed.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a minimally invasive alternative to esophagectomy for early esophageal squamous cell carcinoma (EESCC).The aim of this study was to compare the efficacy and safety of ESD and esophagectomy in EESCC，The data of EESCC patients who received ESD or esophagectomy were retrospectively analyzed. Overall survival (OS), disease specific survival (DSS), recurrence free survival (RFS), and procedure-related variables were compared between ESD and esophagectomy patients.Risk factors affecting the prognosis of patients with early esophageal squamous cell carcinoma were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Mucosal or submucosal squamous cell carcinoma of the esophagus
2. no lymph node involvement or distant metastasis on computed tomography (CT) or pathology;

Exclusion Criteria:

1. Tis premalignant lesions (high-grade intraepithelial neoplasia;HGIN)
2. patients with neoadjuvant therapy
3. patients combined with severe diseases of other organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with early esophageal cancer from January 2011 to January 2021 admitted to Changhai Hospital were included in this study.Patients treated with ESD were classified as the ESD group, and those who underwent radical esophageal cancer treatment were classified as the surgical group.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | 10 years
  OS was measured from the date of ESD or esophagectomy until death from any cause
Disease specific survival (DSS) | 10 years
  DSS was measured from the date of ESD or esophagectomy until death resulting from ESCC
Recurrence free survival (RFS) | 10 years
  RFS was measured from the date of ESD or esophagectomy until the first recurrence or metastasis

SECONDARY OUTCOMES:
postoperative complications | 30 days
  Major postoperative complications includes bleeding, infection, and perforation，stricture and anastomotic leakage, adverse events assessed by blood tests, imageological examination and Endoscopic evaluation. Complications were graded according to the Clavien-Dindo classification system. The higher the complication grade, the more serious.
R0 resection | 15 days
  R0 resection was defined as horizontal and vertical margins free from both cancerous and precancerous tissues (HGIN), and without evidence of LVI. Pathological assessment was performed independently by two pathologists.
adjuvant therapy | 10 years
  During follow-up, record whether Adjuvant therapy (i.e., additional endoscopy/surgery, radiotherapy and/or chemotherapy) was administered.
operation time | 12 hours
  Time from start to finish of operation, measured in minutes
Post-operative hospitalization days | 30 days
  Date of discharge minus date of operation,measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Wei An, Doctor, Principal Investigator — Changhai Hospital, Naval Medical University
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Ding H, Chen T, Zhang X, Chen WF, Li Q, Yao L, Korrapati P, Jin XJ, Zhang YX, Xu MD, Zhou PH. Outcomes of Endoscopic Submucosal Dissection vs Esophagectomy for T1 Esophageal Squamous Cell Carcinoma in a Real-World Cohort. Clin Gastroenterol Hepatol. 2019 Jan;17(1):73-81.e3. doi: 10.1016/j.cgh.2018.04.038. Epub 2018 Apr 25. PMID 29704682
- [Background] An W, Liu MY, Zhang J, Cui YP, Gao J, Wang LP, Chen Y, Yang LX, Chen HZ, Jin H, Liu F, Chen J, Li ZS, Wang LW, Shi XG, Sun C. Endoscopic submucosal dissection versus esophagectomy for early esophageal squamous cell carcinoma with tumor invasion to different depths. Am J Cancer Res. 2020 Sep 1;10(9):2977-2992. eCollection 2020. PMID 33042630
- [Background] Liu Z, Zhao R. Endoscopic Submucosal Dissection vs. Surgery for Superficial Esophageal Squamous Cancer: A Systematic Review and Meta-Analysis. Front Oncol. 2022 Apr 21;12:816832. doi: 10.3389/fonc.2022.816832. eCollection 2022. PMID 35530330
- [Background] Qian M, Feng S, Zhou H, Chen L, Wang S, Zhang K. Endoscopic submucosal dissection versus esophagectomy for t1 esophageal squamous cell carcinoma: a propensity score-matched analysis. Therap Adv Gastroenterol. 2022 Nov 21;15:17562848221138156. doi: 10.1177/17562848221138156. eCollection 2022. PMID 36458047